CLINICAL TRIAL: NCT02810353
Title: Analysis of the Dentoskeletal Effects of the Expander With Differential Opening: a Randomized Clinical Trial
Brief Title: Analysis of the Dentoskeletal Effects of the Expander With Differential Opening
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Arthur César de Medeiros Alves, University of São Paulo, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Bauru Dental School, USP
Record Dates: First submitted 2016-06-18; First posted 2016-06-22 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Maxillary Constriction; Unilateral Posterior Crossbite; Bilateral Posterior Crossbite; Mandibular Dental Arch Constriction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Expander with differential opening group (Experimental): The experimental group will comprise 25 patients who will be submitted to rapid maxillary expansion using the expander with differential opening. The expander will be composed by two 11-mm screws, one anteriorly and the other posteriorly positioned on the palate (Great lakes Orthodontics Ltd, NY, EUA).
  Interventions: Device: Differential rapid maxillary expansion
- Hyrax group (Active Comparator): The control group will be comprised by 25 patients who will undergo rapid maxillary expansion using the conventional Hyrax expander. The expander will be composed by one 11-mm screw centrally positioned on the palate (Dentaurum, Ispringen, Germany).
  Interventions: Device: Conventional rapid maxillary expansion

INTERVENTIONS:
Device: Differential rapid maxillary expansion — Twenty-five patients will be submitted to rapid maxillary expansion using the expander with differential opening. Appliance anchorage will be provided by bands adapted either on the maxillary first permanent molars or on the second deciduous molars and circumferential clamps will be bonded to the maxillary deciduous canines. If the maxillary second deciduous molars will be banded, a lingual extension wire will be placed in the partially erupted maxillary first permanent molars. Both anterior and posterior screws will be activated with a complete turn a day during 6 days. Then, only the anterior screw will be additionally activated for 4 more days. After the active period of RME, the screws will be fixed with acrylic resin and the appliance will be kept as a retainer for 6 months.
  Other Names: RME with the expander with differential opening
  Arms: Expander with differential opening group
Device: Conventional rapid maxillary expansion — Twenty-five patients will undergo rapid maxillary expansion using conventional Hyrax expander. Bands will be adapted either on the maxillary first permanent molars or on second deciduous molars and circumferential clamps will be bonded to the maxillary deciduous canines. Similarly to the experimental group, a lingual extension wire will be placed in the partially erupted maxillary first permanent molars if the maxillary second deciduous molars will be banded. The expander screw will be activated with a complete turn a day during 6 days. After the expansion active phase, the screw will be fixed with acrylic resin and the appliance will be kept in the dental arch as a retainer for 6 months.
  Other Names: RME with the conventional Hyrax expander
  Arms: Hyrax group

SUMMARY:
This study evaluates the dentoskeletal effects of the expander with differential opening in orthodontic patients in the mixed dentition. Half of participants will undergo rapid maxillary expansion (RME) using the expander with differential opening, while the other half will undergo RME using the conventional Hyrax expander.

DETAILED DESCRIPTION:
Recently, a rapid maxillary expander with differential opening was developed aiming to treat maxillary constrictions greater in the anterior region compared to the posterior region of the maxillary dental arch. The aim of this study is to evaluate the dentoskeletal effects of the expander with differential opening in orthodontic patients in the mixed dentition. Material and methods: Fifty patients with maxillary constriction in the mixed dentition will be prospectively and randomly allocated in one of two study groups. The experimental group will comprise 25 patients who will be submitted to rapid maxillary expansion with the expander with differential opening. The control group will be comprised by 25 individuals who will undergo rapid maxillary expander with the Hyrax expander. Digital dental models will be acquired immediately pre-expansion (T1) and six months post-expansion (T2). The Orthoanalyzer™ software will be used to measure maxillary and mandibular widths, arches perimeter, arches lengths, palatal depth, and inclinations of maxillary and mandibular canines and permanent first molars. The intergroup and interphase comparisons will be analyzed using t tests and paired t tests, respectively (p<0.05).

ELIGIBILITY:
Inclusion Criteria:

* Both sexes;
* Ages ranging from 7 to 11 years old;
* Mixed dentition;
* Maxillary constriction;
* No previous orthodontic treatment.

Exclusion Criteria:

* Cleft lip and palate and associated syndromes;
* Systemic and/or neurological diseases.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-12 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Maxillary and mandibular inter-first permanent molar distances | 6 months
Maxillary and mandibular inter-second deciduous molar distances | 6 months
Maxillary and mandibular inter-first deciduous molar distances | 6 months
Maxillary and mandibular inter-deciduous canine distances | 6 months
Maxillary and mandibular dental arches perimeters | 6 months
Maxillary and mandibular dental arches lengths | 6 months
Palatal depth | 6 months
Inclination of maxillary and mandibular first permanent molars | 6 months
Inclination of maxillary and mandibular deciduous canines | 6 months
Amount of interincisor diastema | 10 days

SECONDARY OUTCOMES:
Amount of differential expansion on the maxillary and mandibular dental arches | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Alves, DDS, MSc, Principal Investigator — Bauru Dental School, University of São Paulo
Locations (1):
- University of São Paulo, Bauru, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No